CLINICAL TRIAL: NCT03564509
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group, Dose-range Trial to Investigate the Efficacy and Safety of FE 999302 as add-on Treatment to Follitropin Delta (REKOVELLE) in Women Undergoing Controlled Ovarian Stimulation in a Long GnRH Agonist Protocol
Brief Title: A Trial to Investigate the Efficacy and Safety of FE 999302 as add-on Treatment to Follitropin Delta (REKOVELLE) in Women Undergoing Controlled Ovarian Stimulation.
Acronym: RAINBOW
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000289; 2017-003810-13 (EudraCT Number)
Record Dates: First submitted 2018-05-16; First posted 2018-06-21 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2020-01

CONDITIONS: Controlled Ovarian Stimulation
Keywords: Human Chorionic Gonadotropin (hCG); Recombinant Human Chorionic Gonadotropin (rhCG); Controlled Ovarian Stimulation (COS); Assisted Reproductive Technologies (ART)
MeSH Terms: interventions — follitropin delta; Chorionic Gonadotropin, beta Subunit, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: FE 999302 and placebo were identical in appearance and the trial was considered double-blind as neither the subject nor the investigator knew whether the subject was receiving FE 999302 or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- FE 999302 (1 μg) and follitropin delta (Experimental)
  Interventions: Drug: FE 999302 (1 μg) and follitropin delta
- FE 999302 (2 μg) and follitropin delta (Experimental)
  Interventions: Drug: FE 999302 (2 μg) and follitropin delta
- FE 999302 (4 μg) and follitropin delta (Experimental)
  Interventions: Drug: FE 999302 (4 μg) and follitropin delta
- FE 999302 (8 μg) and follitropin delta (Experimental)
  Interventions: Drug: FE 999302 (8 μg) and follitropin delta
- FE 999302 (12 μg) and follitropin delta (Experimental)
  Interventions: Drug: FE 999302 (12 μg) and follitropin delta
- Placebo and follitropin delta (Placebo Comparator)
  Interventions: Other: Placebo and follitropin delta

INTERVENTIONS:
Drug: FE 999302 (1 μg) and follitropin delta — Daily dose of 1 μg of FE 999302, a recombinant human chorionic gonadotropin (rhCG) solution for subcutaneous injection; individualized follitropin delta dose.
  Other Names: Choriogonadotropin beta
  Arms: FE 999302 (1 μg) and follitropin delta
Drug: FE 999302 (2 μg) and follitropin delta — Daily dose of 2 μg of FE 999302, a rhCG solution for subcutaneous injection; individualized follitropin delta dose.
  Other Names: Choriogonadotropin beta
  Arms: FE 999302 (2 μg) and follitropin delta
Drug: FE 999302 (4 μg) and follitropin delta — Daily dose of 4 μg of FE 999302, a rhCG solution for subcutaneous injection; individualized follitropin delta dose.
  Other Names: Choriogonadotropin beta
  Arms: FE 999302 (4 μg) and follitropin delta
Drug: FE 999302 (8 μg) and follitropin delta — Daily dose of 8 μg of FE 999302, a rhCG solution for subcutaneous injection; individualized follitropin delta dose.
  Other Names: Choriogonadotropin beta
  Arms: FE 999302 (8 μg) and follitropin delta
Drug: FE 999302 (12 μg) and follitropin delta — Daily dose of 12 μg of FE 999302, a rhCG solution for subcutaneous injection; individualized follitropin delta dose.
  Other Names: Choriogonadotropin beta
  Arms: FE 999302 (12 μg) and follitropin delta
Other: Placebo and follitropin delta — Daily dose of placebo; individualized follitropin delta dose.
  Arms: Placebo and follitropin delta

SUMMARY:
The purpose of this phase 2 dose-ranging trial is to investigate the effects of FE 999302 on parameters influencing pregnancy rates in women undergoing Controlled Ovarian Stimulation (COS) with follitropin delta in a long gonadotropin releasing hormone (GnRH) agonist protocol.

Furthermore, the study intends:

* To investigate the safety of FE 999302 in women undergoing COS with follitropin delta in a long GnRH agonist protocol.
* To investigate the potential immunogenicity of FE 999302 in subjects undergoing COS with follitropin delta in a long GnRH agonist protocol.
* To estimate the impact of body weight on FE 999302 exposure in subjects undergoing COS with follitropin delta in a long GnRH agonist protocol.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent documents signed prior to screening evaluations.
* In good physical and mental health as judged by the investigator.
* Anti-Müllerian hormone (AMH) levels at screening of 5.0-35.0 pmol/L (as measured by Elecsys® AMH Plus Immunoassay [Roche Diagnostics] at central laboratory).
* Pre-menopausal women between the ages of 30 and 42 years. The subjects must be at least 30 years (including the 30th birthday) and no more than 42 years (up to the day before the 43rd birthday) when they sign the informed consent.
* Infertile women diagnosed with tubal infertility, unexplained infertility, endometriosis stage I/II or with partners diagnosed with male factor infertility, eligible for in vitro fertilisation and/or intracytoplasmic sperm injection using fresh or frozen ejaculated sperm from male partner or sperm donor.
* Infertility for at least 1 year before screening for subjects less than 35 years or for at least 6 months for subjects greater than equal to (≥)35 years (not applicable in case of tubal or severe male factor infertility).

Exclusion Criteria:

* Known polycystic ovary syndrome (PCOS) associated with anovulation or known endometriosis stage III-IV (defined by the revised American Society for Reproductive Medicine [ASRM] classification, 1996).
* One or more follicles ≥10 mm (including cysts) observed on the transvaginal ultrasound after down-regulation prior to randomisation on stimulation day 1 (puncture of cysts is allowed prior to randomisation).
* Pregnancy (negative pregnancy tests must be documented at screening and prior to start of down-regulation) or contraindication to pregnancy.

Ages: 30 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pre-menopausal women between the ages of 30 and 42 years.
Enrollment: 620 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Number of good-quality blastocysts on Day 5 after oocyte retrieval | On Day 5 after oocyte retrieval
  Quality of blastocysts was assessed by blastocyst expansion and hatching status, blastocyst inner cell mass grading, and trophectoderm grading. The scoring was based on the classification system by Gardner and Schoolcraft, with additional categories for inner cell mass (degenerative or no inner cell mass) and trophectoderm (degenerative or very large cell).

SECONDARY OUTCOMES:
Number of subjects with at least one good-quality blastocyst on Day 5 after oocyte retrieval | On Day 5 after oocyte retrieval
  Quality of blastocysts was assessed by blastocyst expansion and hatching status, blastocyst inner cell mass grading, and trophectoderm grading. The scoring was based on the classification system by Gardner and Schoolcraft, with additional categories for inner cell mass (degenerative or no inner cell mass) and trophectoderm (degenerative or very large cell).
Number of subjects with at least two good-quality blastocysts on Day 5 after oocyte retrieval | On Day 5 after oocyte retrieval
  Quality of blastocysts was assessed by blastocyst expansion and hatching status, blastocyst inner cell mass grading, and trophectoderm grading. The scoring was based on the classification system by Gardner and Schoolcraft, with additional categories for inner cell mass (degenerative or no inner cell mass) and trophectoderm (degenerative or very large cell).
Number and quality of embryos on Day 3 after oocyte retrieval | On Day 3 after oocyte retrieval
  Embryo quality was assessed by cleavage stage and embryo morphology parameters. The total number of embryos and the number of embryos per quality category were reported.
Number and quality of blastocysts on Day 5 after oocyte retrieval | On Day 5 after oocyte retrieval
  Blastocyst quality was assessed by blastocyst expansion and hatching status, blastocyst inner cell mass grading, and trophectoderm grading. The scoring was based on the classification system by Gardner and Schoolcraft, with additional categories for inner cell mass (degenerative or no inner cell mass) and trophectoderm (degenerative or very large cells).
  The total number of blastocysts and the number of blastocysts per quality category will be reported.
Changes in serum hormone levels | Stimulation Day 1 (baseline), stimulation Day 6, stimulation Day 8, end-of-stimulation (up to 20 stimulation days), and oocyte retrieval
  Blood samples for analysis of hormone concentrations were drawn at stimulation Day 1, stimulation Day 6, stimulation Day 8, last day of stimulation, and at oocyte retrieval.
Number and size of follicles on stimulation Day 6 | On stimulation Day 6
  Number and size of follicles assessed using transvaginal ultrasound. The total number of follicles and the number of follicles per size category were reported.
Number and size of follicles at end-of-stimulation | At end-of-stimulation (up to 20 stimulation days)
  Number and size of follicles assessed using transvaginal ultrasound. The total number of follicles and the number of follicles per size category were reported.
Positive beta human chorionic gonadotropin (βhCG) rate | 13-15 days after blastocyst transfer
  Proportion of patients with positive blood βhCG confirmed by a blood test.
Clinical pregnancy rate | 5-6 weeks after blastocyst transfer
  Clinical pregnancy was defined as at least one gestational sac, either intrauterine or ectopic.
Vital pregnancy rate | 5-6 weeks after blastocyst transfer
  Vital pregnancy was defined as at least one intrauterine gestational sac with fetal heart beat, as assessed by transvaginal ultrasound.
Ongoing pregnancy rate | 10-11 weeks after blastocyst transfer
  Ongoing pregnancy was defined as at least one intrauterine viable fetus, assessed using transvaginal or abdominal ultrasound.
Number of oocytes retrieved | On the day of oocyte retrieval
Number of metaphase II oocytes | On the day of oocyte retrieval
Number of fertilised 2 pronuclei (2PN) oocytes | On day 1 after insemination
Total gonadotropin dose | At end-of-stimulation (up to 20 stimulation days)
  The daily dose of FE 999302 or placebo, and follitropin delta were recorded.
Total number of stimulation days | At end-of-stimulation (up to 20 stimulation days)
  The start and end dates of administration of FE 999302 or placebo, and follitropin delta were recorded.
Incidence of cycle cancellation | At end-of-stimulation (up to 20 stimulation days)
  Cycle cancellation due to poor ovarian response or excessive ovarian response.
Serum concentrations of FE 999302 | On stimulation Day 1 (prior to first dose of FE 999302 or placebo), stimulation Day 6, stimulation Day 8, end-of-stimulation (up to 20 stimulation days)
Incidence of ovarian hyperstimulation syndrome (OHSS) (early or late, any grade) | From stimulation Day 1 to end-of-trial (estimated maximum of 4 months from start of stimulation)
  Early OHSS was defined as OHSS with onset less than equal to 9 days after triggering of final follicular maturation.
  Late OHSS was defined as OHSS with onset greater than 9 days after triggering of final follicular maturation.
  All OHSS cases were graded as mild, moderate or severe.
Incidence and intensity of adverse events (AEs) | From screening to end-of-trial (estimated maximum of 4 months from start of stimulation)
Changes in circulating levels of clinical chemistry and haematology parameters | At screening, on stimulation Day 1, end-of-stimulation (up to 20 stimulation days), end-of-trial (estimated maximum of 4 months from start of stimulation)
Incidence and intensity of injection site reactions after FE 999302 administration (redness, pain, itching, swelling and bruising) assessed by the subject during the stimulation period | Immediately after injection of FE 999302 or placebo, 30 minutes after injection, and 24 hours after injection
Incidence of treatment-induced anti-FE 999302 antibodies, overall as well as with neutralising capacity | On stimulation Day 1, end-of-stimulation (up to 20 stimulation days), 19-28 days after the last FE999302 or placebo dose
  The proportion of subjects with treatment-induced anti-FE999302 antibodies as well as the proportion of subjects with treatment-induced anti-FE999302 antibodies with neutralizing capacity were reported.
Incidence of multi-fetal gestation | 5 to 6 weeks after transfer
Incidence of biochemical pregnancy | Up to 5 to 6 weeks after transfer
  Biochemical pregnancy was defined as positive βhCG test but no gestational sac was observed on transvaginal ultrasound conducted later, or menstruation is
  was reported.
Incidence of spontaneous abortion (with and without medical/surgical intervention) | Up to 10 to 11 weeks after transfer
  Spontaneous abortion was defined as positive βhCG test but all intrauterine gestational sacs without fetal heart beat as documented by ultrasound, or there were no viable fetuses observed by ultrasound.
Incidence of ectopic pregnancy (with and without medical/surgical intervention) | Up to 5 to 6 weeks after transfer
  Ectopic pregnancy was defined as extrauterine gestational sac with or without fetal heart beat as documented by ultrasound or surgery.
Incidence of vanishing twins | Up to 10 to 11 weeks after transfer
  Vanishing twin was defined as spontaneous disappearance of an intrauterine gestational sac with or without heart beat in a pregnancy where one viable fetus remained as documented by ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (20):
- Belgium (2):
  - Universitair Ziekenhuis Gent (UZ Gent), Ghent
  - Universitair Ziekenhuis Brussel, Jette
- Czechia (4):
  - Institut fur Reproduktionsmedizin und Genetik, Karlovy Vary
  - Fertimed, Olomouc
  - GYNEM, Prague
  - IVF CUBE, Prague
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Dansk Fertilitetsklinik, Frederiksberg
  - Hvidovre Hospital, Hvidovre
- Spain (6):
  - Dexeus Woman's Health, Barcelona
  - Instituto Valenciano de Infertilidad (IVI) - Bilbao, Leioa
  - GINEFIV - Clinica Belen Location, Madrid
  - Instituto Valenciano de Infertilidad (IVI) - Madrid, Madrid
  - Instituto Valenciano de Infertilidad (IVI) - Sevilla, Seville
  - Instituto Valenciano de Infertilidad (IVI) - Valencia, Valencia
- United Kingdom (4):
  - Glasgow Royal Infirmary, Glasgow
  - Liverpool Women's Hospital, Liverpool
  - Guy's and St Thomas' NHS Trust, London
  - Kings College (Assisted Conception Unit), London

REFERENCES:
- [Result] Sanchez MF, Larsson P, Serrano MF, Bosch E, Velasco JAG, Lopez ES, Mannaerts B. Live birth rates following individualized dosing algorithm of follitropin delta in a long GnRH agonist protocol. Reprod Biol Endocrinol. 2023 May 16;21(1):45. doi: 10.1186/s12958-023-01090-w. PMID 37194068